CLINICAL TRIAL: NCT01098799
Title: Urotensin II in Chronic Kidney Diseases
Brief Title: Urotensin II in Chronic Kidney Diseases and Kidney Transplants
Status: Completed | Type: Observational
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Hursitoglu, Chair, Vakif Gureba Training and Research Hospital
Other Study IDs: Dahiliye-2-Urotensin
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Renal Disease
Keywords: Urotensin II,Chronic renal disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Healthy controls
- Chronic kidney disease-1: Chronic kidney disease not taking dialysis treatment
- Kidney Transplant: Kidney transplants

SUMMARY:
The investigators are planning to study the serum level of Urotensin II in chronic kidney disease patients, kidney transplants, and healthy controls.

DETAILED DESCRIPTION:
The investigators will determine the urotensin II levels in Chronic kidney disease patients, kidney transplants, and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18

Exclusion Criteria:

* Inability to give a written consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls,CRF patients and kidney transplants aged more than 18
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
serum Urotensin II(UII)level | at enrollment
  We tried to compare UII level in normal, chronic kidney disease and kidney transplant patients group

CONTACTS AND LOCATIONS:
Overall Officials: Tufan Tukek, MD, Study Director — Vakif Gureba Training & Research Hospital
Locations (1):
- Vakif Gureba Training & Research Hospital, Istanbul, Turkey (Türkiye)